CLINICAL TRIAL: NCT04399252
Title: A Randomized Trial of the Effect of Lactobacillus on the Microbiome of Household Contacts Exposed to COVID-19
Brief Title: Effect of Lactobacillus on the Microbiome of Household Contacts Exposed to COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro00105674
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Microbiome
Keywords: COVID-19; Lactobacillus rhmanosus GG
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LGG Arm (Experimental): Participants in this arm will be given LGG for 28 days.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG
- Placebo (Placebo Comparator): Participants in this arm will be given a placebo for 28 days.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG — Participants will take 2 capsules per day of either LGG or placebo.
  Arms: LGG Arm
Dietary Supplement: Lactobacillus rhamnosus GG Placebo — Participants will take 2 capsules per day of LGG placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of the probiotic Lactobacillus rhamnosus GG (LGG) and the effect of COVID-19 on the microbiome (the microorganisms that live in and on the human body) in exposed household contacts of COVID-19. This is a randomized, double-blind, placebo-controlled study, meaning subjects will be randomly assigned to receive LGG or a placebo (an inactive substance given in the same form as the active substance) and will not know which product they are receiving. Subjects will participate in the study for around 60 days. All subjects must refrain from taking any other probiotics while on study. All subjects must have access to e-mail and the internet to complete study questionnaires. Participation in this study entails taking LGG/placebo for 28 days, responding to questionnaires, and providing stool and nasal swab samples.

ELIGIBILITY:
Inclusion Criteria:

* Age >=1 year (as children <1 year may not be able to take oral probiotics)
* Household contact of someone diagnosed with COVID-19
* Willingness to stop taking other probiotics or to not take any other probiotic while on LGG/placebo (taking a probiotic at the time of screening will not be considered a reason for exclusion. However, subjects will be asked to stop taking their probiotic if they enroll on the study).
* Access to e-mail/internet to complete electronic consent via REDCap

Exclusion Criteria:

* Symptoms of COVID-19 at enrollment, including:

  * Fever
  * Respiratory symptoms
  * GI symptoms
  * Anosmia
  * Ageusia ->7 days since original patient associated with household contact was diagnosed with COVID-19
* Taking hydroxychloroquine or remdesivir for any reason (as this would have the potential to decrease the expected rate of COVID-19 in this population and affect our power and sample size calculations)
* Enrolled in a COVID-19 prophylaxis study (as this would have the potential to decrease the expected rate of COVID-19 in this population and affect our power and sample size calculations)
* Any medical condition that would prevent taking oral probiotics or increase risks associated with probiotics including but not limited to:

  * Inability to swallow/aspiration risk and no other methods of delivery (e.g., no G/J tube)
  * Increased infection risk due to immunosuppression due to:

    * Chronic immunosuppressive medication
    * Prior organ or hematopoietic stem cell transplant
    * Known neutropenia (ANC <500 cells/ul)
    * HIV and CD4 <200 cells/ul
  * Increased infection risk due to endovascular due to:

    * Rheumatic heart disease
    * Congenital heart defect,
    * Mechanical heart valves
    * Endocarditis
    * Endovascular grafts
    * Permanent endovascular devices such as permanent (not short-term) hemodialysis catheters, pacemakers, or defibrillators
  * Increased infection risk due to mucosal gastrointestinal due to:

    * Gastroesophageal or intestinal injury, including active bleeding

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of one or more symptoms of COVID-19 during the study period | 60 days
  Incidence of one or more symptoms of COVID-19 (fever, chills, headache, muscle aches, runny nose, sore throat, cough, shortness of breath, nausea or vomiting, diarrhea, stomach upset or pain, excessive bloating or gas, constipation, loss of sense of smell, loss of sense of taste, rash, painful toes, or other symptoms related to COVID-19 diagnosis) during the study period

SECONDARY OUTCOMES:
Incidence of laboratory-confirmed COVID-19 during the study period | 60 days
  Incidence of laboratory-confirmed COVID-19 (all based on medically-dictated, clinical testing and electronic medical record review) or research laboratory-confirmed COVID-19 (all, based on research testing of nasal swab and stool samples) during the study period
Complications of COVID-19 | 60 days
  Complications of COVID-19 (e.g., need for hospitalization, intubation, mortality) during the study period
Types of symptoms of COVID-19 | 60 days
  Types of symptoms of COVID-19 during the study period (e.g., fever, chills, headache, muscle aches, runny nose, sore throat, cough, shortness of breath, nausea or vomiting, diarrhea, stomach upset or pain, excessive bloating or gas, constipation, loss of sense of smell, loss of sense of taste, rash, painful toes, or other symptoms related to COVID-19 diagnosis)
Duration of symptoms of COVID-19 | 60 days
  Duration of symptoms (days) of COVID-19 during the study period

OTHER OUTCOMES:
Change in Shannon Diversity in patients that develop COVID-19 | Baseline, Day 7, Day 28
  Impact of COVID-19 on and of the microbiome, as determined by Shannon Diversity of stool and nasal swab samples, during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sung, MD, Principal Investigator — Duke University; Paul Wischmeyer, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wischmeyer PE, Tang H, Ren Y, Bohannon L, Jiang D, Bergens M, Ramirez ZE, Andermann TM, Messina JA, Sung JA, Jensen D, Jung SH, Artica A, Britt A, Bush A, Johnson E, Lew MV, Winthrop H, Pamanes C, Racioppi A, Zhao AT, Wan Z, Surana NK, Sung AD. Efficacy of probiotic treatment as post-exposure prophylaxis for COVID-19: A double-blind, Placebo-Controlled Randomized trial. Clin Nutr. 2024 Jan;43(1):259-267. doi: 10.1016/j.clnu.2023.11.043. Epub 2023 Dec 11. PMID 38103462
- [Derived] Tang H, Bohannon L, Lew M, Jensen D, Jung SH, Zhao A, Sung AD, Wischmeyer PE. Randomised, double-blind, placebo-controlled trial of Probiotics To Eliminate COVID-19 Transmission in Exposed Household Contacts (PROTECT-EHC): a clinical trial protocol. BMJ Open. 2021 May 5;11(5):e047069. doi: 10.1136/bmjopen-2020-047069. PMID 33952552
- See also: Pre-print: Daily Lactobacillus Probiotic versus Placebo in COVID-19-Exposed Household Contacts (PROTECT-EHC): A Randomized Clinical Trial — https://www.medrxiv.org/content/10.1101/2022.01.04.21268275v1